CLINICAL TRIAL: NCT04965896
Title: The Effect of Nut Intake At Night on Postprandial Glycaemia: a Randomised Crossover Trial in Healthy Adults
Brief Title: Nut Intake At Night: Effect on Postprandial Glycaemia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Trial was planned for 2020, but Melbourne 2020 and 2021 lockdowns hindered the study.
Sponsor: Monash University (Other)
Responsible Party: Principal Investigator, Barbara R. Cardoso, Lecturer, Monash University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Nut-night glucose response
Record Dates: First submitted 2021-07-08; First posted 2021-07-16 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Postprandial Hyperglycemia; Insulin Resistance
Keywords: glucose tolerance; meal timing; insulin; nuts; postprandial
MeSH Terms: conditions — Hyperglycemia; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Participants will complete 2 study sessions at night, consuming plain white rice (corresponding to 75g of available carbohydrate) alongside each test meal (either the nuts or control meal) on two separate occasions. The order of scheduling of the sessions will be randomised.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control meal (Placebo Comparator): Participants will receive plain white rice (75g of available carbohydrate) alongside a snack with crackers and cheese. The meal is similar in energy and macronutrients to the test meal.
  Interventions: Other: Control meal
- Nut meal (Experimental): Participants will receive plain white rice (75g of available carbohydrate) alongside a portion of 30g of nuts. The meal is similar in energy and macronutrients to the control meal.
  Interventions: Other: Nut meal

INTERVENTIONS:
Other: Control meal — Participants will receive plain white rice (75g of available carbohydrate) alongside a snack with crackers and cheese. The meal is similar in energy and macronutrients to the test meal.
  Arms: Control meal
Other: Nut meal — Participants will receive plain white rice (75g of available carbohydrate) alongside a portion of 30g of nuts. The meal is similar in energy and macronutrients to the control meal.
  Arms: Nut meal

SUMMARY:
There is some evidence to suggest that the timing of a meal intake directly impacts postprandial insulin and glucose responses, with meals consumed later during the day being more metabolically detrimental that the same meals consumed during the day. This information is particularly pertinent to the 16% of people employed in shift-work professions in Australia who have little choice but to eat during the late evening and overnight. The purpose of this study is to compare two effect of different meals or snacks (control vs test meal) on blood glucose and insulin at night time in healthy adults. This study will enable to develop suitable meals to consume at night time that can reduce the higher glucose and insulin responses that are a consequence of eating late into the night.

DETAILED DESCRIPTION:
Eating in the morning results in a more effective clearance of blood sugar (glucose). However, some people, such as shift workers, have no choice but to eat at night. Previous studies have shown that consuming protein at night can be effective at lowering blood sugar. The investigators here propose that nuts would be a healthy snack to eat at night time as they are a good source of protein and may help to reduce the high levels of blood glucose observed by eating at night time.

The aim of this cross-over study is to compare the effect of a snack high in nuts compared with a control snack similar in macronutrients (cheese and crackers) on postprandial blood glucose and insulin in healthy participants after consumption of a meal known to raise blood sugar (white rice). The investigators hypothesise that compared with a standard snack, a snack containing nuts will show a lower postprandial glucose and insulin response.

The participants will complete an initial screening questionnaire to check eligibility. Eligible participants will attend the research facilities after 5h fasting at night (from 18.30pm-22.00pm) on two occasions, when they will receive plain white rice (75g of available carbohydrate) alongside either 30 g of mixed nuts (test meal) or a snack with cheese and crackers (control meal) that is equivalent in energy and macronutrient content. During the visits, a finger prick fasting glucose sample will be collected. Repeated finger prick samples will be collected at 15, 30, 45, 60, 90, 120, 150 and 180 minutes after the meal intake. These samples will be used for glucose and insulin measurement. Postprandial glucose and insulin iAUC will be calculated. Differences in glucose and insulin concentrations and iAUC as well as glucose time to peak will be compared between the two treatment conditions.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 50 years of age
* Waist circumference of <94cm and <80cm for Caucasian males and females, respectively
* Waist circumference of <90cm and <80 cm for Asian males and females, respectively
* Available to attend two testing sessions at the research facility

Exclusion Criteria:

* Diagnosed with type 2 diabetes or taking anti-diabetic medication (oral hypoglycaemic agents)
* Impaired fasting glucose (≥ 7 mmol/L)
* Gastrointestinal conditions that may affect glycaemic response
* Serious health conditions that may affect participation e.g. liver or thyroid dysfunction, recent major surgery
* Women planning pregnancy, pregnant or lactating.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Postprandial plasma glucose area under the curve (iAUC) | Three hour glucose iAUC will be calculated at nine time points (0, 15, 30, 45, 60, 90, 120, 150 and 180 mins) after beginning consumption of the test meal.
  Difference in postprandial plasma glucose iAUC
Postprandial plasma insulin iAUC | Three hour glucose iAUC will be calculated at seven time points (0, 30, 60, 90, 120, 150 and 180 mins) after beginning consumption of the test meal.
  Difference in postprandial plasma insulin iAUC

SECONDARY OUTCOMES:
Postprandial glucose concentration | Glucose concentration will be measured at nine time points (0, 15, 30, 45, 60, 90, 120, 150 and 180 mins) after beginning consumption of the test meal.
  Difference in postprandial glucose concentration
Postprandial insulin concentration | Insulin concentration will be measured in finger prick blood samples at seven time points (0, 30, 60, 90, 120, 150 and 180 mins) after beginning consumption of the test meal.
  Difference in postprandial insulin concentration
Time to peak glucose | Three hours
  Difference in time to peak glucose

IPD SHARING:
Plan to Share IPD: No